CLINICAL TRIAL: NCT02399059
Title: Effect of Peritoneal Lavage With Clindamycin-Gentamicin Solution During Elective Colorectal Cancer Surgery on the Oncologic Outcome
Brief Title: Effect of Peritoneal Lavage With Clindamycin-Gentamicin Solution & Oncologic Outcome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, MD, PhD, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HURJ2015-01
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Colorectal Tumors
Keywords: recurrence
MeSH Terms: conditions — Colorectal Neoplasms; Recurrence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antibiotic lavage (Experimental): Peritoneal irrigation with Gentamycin - clndamycin solution
  Interventions: Procedure: Antibiotic lavage
- Normal saline lavage (Active Comparator): Peritoneal irrigation with normal saline
  Interventions: Procedure: Normal saline lavage

INTERVENTIONS:
Procedure: Antibiotic lavage — Peritoneal irrigation with gentamycin-clindamycin solution
  Arms: Antibiotic lavage
Procedure: Normal saline lavage — Peritoneal irrigation with normal saline
  Arms: Normal saline lavage

SUMMARY:
Antibiotic lavage reduces bacterial contamination and decreases SSI infection rate. SSI leads to an immunocompromised situation, leaving unattended the neoplasm. It has been described that SSI may result in a worse oncologic outcome.

DETAILED DESCRIPTION:
Antibiotics combined with lavage have demonstrated a reduction in the bacterial contamination and decreases SSI infection rate. SSI leads to an immunocompromised situation, as immunologic defense is focused on controlling the septic focus, leaving unattended the neoplasm. It has been described that SSI may result in a worse oncologic outcome. The aim of this study is to evaluate prospectively the effect of peritoneal lavage with clindamycin and gentamicin on the oncologic outcome of colorectal tumours.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of colon neoplasms
* plans to undergo an elective surgery with curative aims

Exclusion Criteria:

* preoperative diagnosis of chronic renal failure (because of the risk of nephrotoxicity associated with intraperitoneal gentamicin absorption)
* allergy to gentamicin or clindamycin.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2011-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Global survival | 36 months after intervention

SECONDARY OUTCOMES:
Disease free survival | 36 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Ruiz-Tovar, MD, PhD, Principal Investigator — Hospital Rey Juan Carlos